CLINICAL TRIAL: NCT03109080
Title: A Phase I of Olaparib With Radiation Therapy in Patients With Inflammatory, Loco-regionally Advanced or Metastatic TNBC (Triple Negative Breast Cancer) or Patient With Operated TNBC With Residual Disease
Brief Title: Olaparib & Radiation Therapy for Patients Triple Negative Breast Cancer (TNBC)
Acronym: RadioPARP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2016-01 RadioPARP; 2016-001837-28 (EudraCT Number)
Record Dates: First submitted 2017-03-02; First posted 2017-04-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasms, Triple-Negative; Breast Neoplasm Malignant Female; Radiotherapy Side Effect
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Radiation Injuries | interventions — olaparib; Poly A; Adenosine Diphosphate; Adenosine Diphosphate Ribose; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib + radiation therapy (Experimental): One week of Olaparib alone followed by 5 weeks of Olaparib and concurrent loco-regional radiotherapy. Five levels of dose of Olaparib are expected.
  Interventions: Drug: Olaparib; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Olaparib — five levels of dose, per os administration, twice daily each day
  Other Names: PARP (Poly (Adenosine diphosphate [ADP]-Ribose) Polymerase) inhibitor, Lynparza, AZD-2281
Radiation: Radiation therapy — 3D conformal radiotherapy or intensity-modulated radiotherapy (IMRT), Simultaneous Integrated Boost (SIB), postoperative radiotherapy
  Other Names: Radiotherapy

SUMMARY:
A Phase I of Olaparib with Radiation Therapy in Patients With Inflammatory, Loco-regionally Advanced or Metastatic TNBC (triple negative breast cancer) or Patient With Operated TNBC with Residual Disease.

DETAILED DESCRIPTION:
Open label phase I, dose escalation trial for patients with triple negative inflammatory, loco-regional advanced or metastatic breast cancer either inoperable after neoadjuvant chemotherapy or operated with residual disease (after neoadjuvant chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

1. Woman aged >18 years.
2. Histologically confirmed triple negative breast cancer with loco-regional radiotherapy indication :

   1. Non-operated with either:

      1. Inflammatory breast cancer in progression during neoadjuvant chemotherapy or inoperable after neoadjuvant chemotherapy.
      2. Loco-regional advanced breast cancer in progression during neoadjuvant chemotherapy or inoperable after neoadjuvant chemotherapy (T ≥ 3 and/or N ≥ 1; with evaluable disease according to RECIST 1.1 criteria).
      3. Non operable metastatic breast cancer (all T, all N, M1; with evaluable disease according to RECIST 1.1 criteria) needing local and regional treatment in case of good metastatic control after chemotherapy.
   2. Or patient operated after neoadjuvant treatment and surgery with residual disease (non-pCR and/or pN+ disease).
3. Neoadjuvant chemotherapy (containing anthracyclines or taxanes or the combination of both or containing platinum-based chemotherapy) willingness to discontinue any cytotoxic chemotherapeutic agents, immunotherapy, and targeted therapies at least two weeks prior to start of Olaparib.
4. ECOG performance status < 2.
5. Life expectancy greater than 6 months.
6. Adequate hematologic, renal and hepatic function (assessed within the two weeks prior to registration and within the month prior to the commencement of protocol treatment). For patients who have stopped chemotherapy two weeks prior to protocol treatment, hematologic function must be re-assessment 1 or 2 days before the first Olaparib intake:

   1. Haemoglobin ≥ 10.0 g/dL.
   2. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L.
   3. White Blood Cells (WBC) > 3 x 109/L.
   4. Platelet count ≥ 100 x 109/L.
   5. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (except in case of Gilbert syndrome).
   6. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5 x ULN.
   7. Patients must have Creatinine Clearance estimated using the Cockcroft-Gault equation of ≥ 51 mL/min
7. Urine or serum negative pregnancy test within two weeks prior to registration for non-postmenopausal patients. Negative pregnancy test confirmed within 1 or 2 days prior to first Olaparib intake.
8. For woman with child-bearing potential, an efficacious contraception following sponsor recommendations must be used during the whole treatment period and up to three months after the last Olaparib administration.
9. Ability to swallow and retain oral medications without gastrointestinal disorders likely to interfere with absorption of the study medication.
10. Affiliation to the French Social Security System.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Radiation therapy: prior history of radiation therapy to the ipsilateral breast and/or regional nodes (except prior radiation therapy to other sites).
2. Patient with unresolved or unstable, NCI-CTCAE v4.03 (National Cancer Institute Common Toxicity Criteria for Adverse Events) Grade 3 or greater toxicity from prior administration of prior anti-cancer treatment.
3. Patient with clinically and uncontrolled significant comorbidity: major cardiac, respiratory, renal, hepatic, gastrointestinal, hematologic or neurological/psychiatric disease or disorder, including but not limited to: active uncontrolled infection; symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia; any other illness condition(s) that could exacerbate potential toxicities, require excluded therapy for management, or limit compliance with study requirements.
4. Patient with second primary cancer, except : adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years.
5. Concomitant anti-cancer treatment during protocol treatment and/or not completed at least 2 weeks prior to Olaparib initiation, except bisphosphonates and RANK inhibitors without restriction even during protocol treatment as long as these where started at least 4 weeks prior to study treatment initiation.
6. Any previous treatment with a PARP (Poly (Adenosine diphosphate [ADP]-Ribose) Polymerase) inhibitor, including Olaparib.
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Olaparib.
8. Patient being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A (Rifabutin, Rifampicin, Clarithromycin, Ketoconazole, Itraconazole, Voriconazole, Ritonavir, Telithromycin) within the last 7 days before first Olaparib intake.
9. Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
10. Blood transfusions within 14 days prior to treatment start.
11. Patient with myelodysplastic syndrome / acute myeloid leukaemia.
12. Pregnant or breastfeeding woman.
13. Patient already included in another clinical trial with an investigational drug.
14. Patient individually deprived of liberty or placed under the authority of a tutor.
15. Patient with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Determination of the Maximal Tolerated Dose of Olaparib administered with concurrent loco regional radiotherapy | 2 years
  Incidence of early Dose Limited Toxicity (DLTs: early adverse effects related to Olaparib administered with concurrent radiotherapy) to determinate the Maximal Tolerated Dose (MTD) of Olaparib administered with concurrent loco regional radiotherapy in patients who have triple negative inflammatory, loco-regional advanced or metastatic breast cancer either inoperable after neoadjuvant chemotherapy or operated patient with residual disease (after neoadjuvant chemotherapy).

SECONDARY OUTCOMES:
Incidence of Serious Adverse Events (SAEs), graded according to NCI-CTCAE version 4.03 criteria to assess the safety profile of Olaparib administered with concurrent loco-regional radiotherapy. | 2 years
  Incidence of Serious Adverse Events (SAEs), graded according to NCI-CTCAE version 4.03 criteria
Incidence and severity of Adverse Events (AEs), graded according to NCI-CTCAE version 4.03 criteria to assess the safety profile of Olaparib administered with concurrent loco-regional radiotherapy. | 2 years
  Incidence and severity of Adverse Events (AEs), graded according to NCI-CTCAE version 4.03 criteria
Incidence and severity of laboratory abnormalities, graded according to NCI-CTCAE version 4.03 criteria to assess the safety profile of Olaparib administered with concurrent loco-regional radiotherapy. | 2 years
  Incidence and severity of laboratory abnormalities, graded according to NCI-CTCAE version 4.03 criteria
Incidence of acute toxicity 2 weeks and 6 weeks after the end of radiotherapy to assess the safety profile of Olaparib administered with concurrent loco-regional radiotherapy. | 2 years
  Incidence of acute toxicity 2 weeks and 6 weeks after the end of radiotherapy
Incidence of late toxicity at 1 year and at 2 years as of initiation of radiation therapy to assess the safety profile of Olaparib administered with concurrent loco-regional radiotherapy. | 2 years
  Incidence of late toxicity at 1 year and at 2 years as of initiation of radiation therapy
Incidence of treatment discontinuations and treatment modifications due to AEs to assess the safety profile of Olaparib administered with concurrent loco-regional radiotherapy. | 2 years
  Incidence of treatment discontinuations and treatment modifications due to AEs
Evaluation of the Objective Response Rate (ORR) to evaluate Olaparib administered with concurrent loco regional radiotherapy efficacy profile | 2 years
  Evaluation of the Objective Response Rate (ORR) to treatment
Evaluation of the Complete Response Rate to evaluate Olaparib administered with concurrent loco regional radiotherapy efficacy profile | 2 years
  Evaluation of the Complete Response Rate to treatment
Evaluation of Pathological Response Rate (pRR) after salvage surgery to evaluate Olaparib administered with concurrent loco regional radiotherapy efficacy profile | 2 years
  Evaluation of Pathological Response Rate (pRR) after salvage surgery
Evaluation of the loco-regional Progression Free Survival (l-PFS) to evaluate Olaparib administered with concurrent loco regional radiotherapy efficacy profile | 2 years
  Evaluation of the loco-regional Progression Free Survival (l-PFS)
Evaluation of the Progression Free Survival (PFS) or Disease Free survival (DFS) according to stage of disease to evaluate patient outcome | 2 years
  Evaluation of the Progression Free Survival (PFS) or Disease Free survival (DFS)
Evaluation of the distant relapse rate to evaluate patient outcome | 2 years
  Evaluation of the distant relapse rate
Evaluation of patient outcome by evaluation of the Overall Survival (OS). | 2 years
  Evaluation Overall Survival (OS).
Evaluation of patient outcome by evaluate disease specific survival rate. | 2 years
  Evaluation of the disease specific survival rate.
Explore biomarkers of Olaparib activity in combination with concurrent radiotherapy. | 2 years
  Exploration of biomarkers of Olaparib associated with radiotherapy on biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Youlia KIROVA, MD, Study Director — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Result] Loap P, Loirat D, Berger F, Ricci F, Vincent-Salomon A, Ezzili C, Mosseri V, Fourquet A, Ezzalfani M, Kirova Y. Combination of Olaparib and Radiation Therapy for Triple Negative Breast Cancer: Preliminary Results of the RADIOPARP Phase 1 Trial. Int J Radiat Oncol Biol Phys. 2021 Feb 1;109(2):436-440. doi: 10.1016/j.ijrobp.2020.09.032. Epub 2020 Sep 21. PMID 32971187
- [Derived] Loap P, Loirat D, Berger F, Rodrigues M, Bazire L, Pierga JY, Vincent-Salomon A, Laki F, Boudali L, Raizonville L, Mosseri V, Jochem A, Eeckhoutte A, Diallo M, Stern MH, Fourquet A, Kirova Y. Concurrent Olaparib and Radiotherapy in Patients With Triple-Negative Breast Cancer: The Phase 1 Olaparib and Radiation Therapy for Triple-Negative Breast Cancer Trial. JAMA Oncol. 2022 Dec 1;8(12):1802-1808. doi: 10.1001/jamaoncol.2022.5074. PMID 36301572